CLINICAL TRIAL: NCT04043390
Title: A One-stop Shop for the Same Day Diagnosis and Management of TB and HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: REACH Ethiopia (Unknown); Bingham University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-063
Record Dates: First submitted 2018-12-19; First posted 2019-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Tuberculosis; Hiv
Keywords: Xpert MTB/RIF; tuberculosis; diagnostics; Xpert Ultra; Truenat MTB; Truenat MTB RIF; C Reactive Protein; Xpert HIV-1 VL; Truenat HIV-1 VL; C Reactive Protein QUBE
MeSH Terms: conditions — Tuberculosis; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: This will be a phase III open randomised diagnostic trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CRP and Xpert ULTRA MTB/RIF (Experimental): Scheme 1 will screen all patients for HIV using rapid tests routinely used by the clinics and a rapid CRP. Patients with CRP >10 will be further tested using Xpert ULTRA. Individuals with HIV will undergo an HIV VL using Xpert HIV-1 VL.
  Interventions: Diagnostic Test: CRP and Xpert ULTRA MTB/RIF; Diagnostic Test: standard test Xpert; Diagnostic Test: Culture as reference standard
- CRP and Molbio Truenat MTB (Experimental): Scheme 2 will screen individuals for HIV and CRP (as in scheme 1) and patients with CRP >10 will be tested using Molbio Truenat MTB. Individuals with HIV will undergo an HIV VL using Molbio Truenat HIV-VL and individuals with Truenat MTB-positive samples wil be tested with Truenat MTB RIF.
  Interventions: Diagnostic Test: CRP and Molbio Truenat MTB; Diagnostic Test: standard test Xpert; Diagnostic Test: Culture as reference standard
- standard test Xpert (No Intervention): All patients receiving in scheme 1 and scheme 2 will be tested using the standard tests used in the study context. These are rapid HIV tests, Xpert MTB/RIF and culture.

INTERVENTIONS:
Diagnostic Test: CRP and Molbio Truenat MTB — A molecular assay to detect M tuberculosis DNA Truenat is currently undergoing the process of endorsement by the WHO.
  Other Names: CRP and Truelab MTB
  Arms: CRP and Molbio Truenat MTB
Diagnostic Test: CRP and Xpert ULTRA MTB/RIF — A molecular assay to detect M tuberculosis DNA ULTRA is already endorsed by the WHO. However the tests are still considered experimental in Nigeria and Ethiopia.
  Other Names: CRP and ULTRA
  Arms: CRP and Xpert ULTRA MTB/RIF
Diagnostic Test: standard test Xpert — The investigators will use Xpert to compare its agreement with scheme 1 (CRP plus Truenat MTB) and scheme 2 (CRP plus ULTRA).
  Arms: CRP and Molbio Truenat MTB; CRP and Xpert ULTRA MTB/RIF
Diagnostic Test: Culture as reference standard — The investigators will use culture to assess the sensitivity of schemes 1 and 2
  Arms: CRP and Molbio Truenat MTB; CRP and Xpert ULTRA MTB/RIF

SUMMARY:
TB is a major public health problem and the second most common cause of adult death due to infection in many low-income countries. Despite major efforts to de-centralise services, accessibility to diagnosis is still limited, with one third of the 9 million cases occurring each year being missed by national control programmes.

New TB diagnostics suitable for use at the point-of-care are emerging. Some of these are intended for screening purposes, as an initial step to identify individuals who may have TB and should undergo further tests for confirmation. These tests may have high sensitivity, but also give false-positive results (low specificity). Other tests aim to be the confirmatory tests for TB (high specificity), but these tests are often more expensive and complex and are only available in hospital laboratories. As these tests have different purposes, it is likely they would work better in combination in a step fashion to optimise their impact and to develop an efficient diagnostic process. Furthermore, as none of the tests is versatile enough to be used in all settings, test combinations will need to consider the health system context in which they would be used. Our aim is to develop and evaluate rapid and accurate diagnostic approaches for TB that facilitate the initiation of appropriate treatment on the same day of the initial consultation in Africa.

The objectives are to

1. Evaluate new diagnostics for TB (including among HIV co-infected individuals) that are suitable at the point-of-care;
2. Develop diagnostic algorithms that streamline and accelerate the diagnosis of TB, allowing patients to reach clinical management decisions within a single clinic visit;
3. Determine the impact of using novel point-of-care diagnostic combinations on the proportion of patients correctly initiating TB treatment within 24-48 hours of first attendance; their potential cost effectiveness

The investigators conducted studies in 2016-2018 to accomplish the first two objectives and have identified diagnostic tests that are suitable for low and middle income countries.

This document therefore refers to objective 3, which aims to

1. Assess the performance of two diagnostic schemes for the diagnosis of TB when compared to culture.
2. Assess the yield of two diagnostic schemes for the diagnosis of TB when compared to Xpert and
3. Assess the cost of the two diagnostic schemes compared to Xpert.

DETAILED DESCRIPTION:
The study will enrol patients in TB clinics based in 4 selected district hospitals (two in Nigeria and two in Ethiopia) and samples will be processed in a single reference laboratory. This diagnostic evaluation trial will comprise two experimental diagnostic schemes which will be compared against the standard of care:

* One experimental arm (scheme 1) will screen all patients for HIV using two rapid tests routinely used by the clinics and a rapid CRP. Selected patients will be further tested using ULTRA. Individuals with HIV will undergo an HIV VL using Xpert.
* A second experimental arm (scheme 2): will screen individuals for HIV and CRP (as in scheme 1) and selected patients will be tested using Molbio Truenat MTB. Individuals with HIV will undergo an HIV VL using Molbio Truenat HIV-VL and Truenat RIF.
* In addition, all patients will be tested using the standard of care consistent of confirmatory HIV and CRP tests, Xpert MTB/RIF and culture.

  * Randomisation All patients will be randomised at a ratio of 1:1 into schemes 1 and 2. Random numbers will be generated in LSTM by a statistician independent to the study. The scheme allocations will be included in study envelopes assigned to individual study numbers. Equal number of participants will be included in Nigeria and Ethiopia.
  * Proposed methods for protecting against source bias

As this is an open trial, the classification of patients will be based on objective quantitative results of laboratory tests. It is expected the test performances will vary according to HIV status. Participants will be classified according to their experimental test results

ELIGIBILITY:
Inclusion Criteria:

1. Adult with presumptive TB
2. At least one of the following criteria: Cough > 2-week duration, weight loss, unexplained fever, night sweats or haemoptysis.
3. Willing to participate in the study

Exclusion Criteria:

1. Age unknown and likely being a minor (looks <18 years old)
2. Known pregnancy
3. Has received or is receiving anti-TB treatment
4. Already diagnosed with TB.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Performance of two diagnostic schemes for the diagnosis of TB when compared to culture. | "up to two months", once culture results become available
  Sensitivity, specificity, positive and negative predictive values of schemes 1 and 2 to identify patients with TB. Culture will used as the reference standard.

SECONDARY OUTCOMES:
Agreement of two diagnostic schemes for the diagnosis of TB when compared to Xpert. | "up to two months", once culture results become available
  Assessment of the agreement between the results obtained with schemes 1 and 2 and Xpert MTB/RIF.
  Xpert MTB/RIF is the recommended test for diagnosis and patients are managed according to their Xpert MTB/RIF results and clinical assessment. The investigators will describe whether the use of the schemes would result in a similar yield than the yield obtained by Xpert.
Time required for diagnosis of the two diagnostic schemes compared to Xpert. | 10 months
  The investigators will describe the time required to achieve a diagnosis.
Cost required for diagnosis of the two diagnostic schemes compared to Xpert. | 10 months
  The investigators will describe the costs of the tests in schemes 1 and 2 and compare these costs with the costs of screening all patients with Xpert MTB/RIF.

CONTACTS AND LOCATIONS:
Overall Officials: Luis E Cuevas, Professor, Principal Investigator — Liverpool School of Tropical Medicine
Locations (1):
- Zankli Research Centre, Kobape, Nasarawa State, Nigeria

IPD SHARING:
Plan to Share IPD: No
Data will be made open access once primary results are published and within 6 months of database lock. Data will be shared with WHO for the purpose of diagnostic endorsement.

REFERENCES:
- [Derived] Inbaraj LR, Daniel J, Sathya Narayanan MK, Srinivasalu VA, Bhaskar A, Scandrett K, Rajendran P, Kirubakaran R, Shewade HD, Malaisamy M, Padmapriyadarsini C, Takwoingi Y. Truenat MTB assays for pulmonary tuberculosis and rifampicin resistance in adults and adolescents. Cochrane Database Syst Rev. 2025 Mar 24;3(3):CD015543. doi: 10.1002/14651858.CD015543.pub2. PMID 40122135